CLINICAL TRIAL: NCT00003812
Title: Topotecan/Paclitaxel Induction Followed by Consolidation Chemoradiotherapy for Limited Stage Small Cell Lung Cancer: A Phase II Study
Brief Title: Chemotherapy Plus Radiation Therapy in Treating Patients With Limited-Stage Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CALGB-39808; U10CA031946 (NIH); CLB-39808; CDR0000066958 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 1999-11-01; First posted 2004-07-22 (Estimated); Last update posted 2016-07-20 (Estimated); Status verified 2016-07

CONDITIONS: Lung Cancer
Keywords: limited stage small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Filgrastim; Carboplatin; Etoposide; Paclitaxel; Topotecan; Radiotherapy

ARMS (1):
- chemotherapy + radiation therapy (Experimental): Patients receive topotecan IV on days 1-5 and paclitaxel IV over 3 hours on day 1. Filgrastim (G-CSF) is administered subcutaneously every day starting on day 6 until blood counts recover. The course is repeated once beginning on day 22. After restaging, patients begin thoracic radiotherapy daily, five days per week, for 6-7 weeks. On the same day that radiotherapy begins, patients receive carboplatin IV over 1 hour (day 43) and etoposide IV over 1 hour daily for 3 days (days 43-45). The consolidation chemotherapy is repeated every 21 days for a total of 3 courses. Patients with stable or responding disease undergo prophylactic cranial irradiation. Patients are followed at least every 3 months for 2 years, every 6 months for 3 years, and then at least every year.
  Interventions: Biological: filgrastim; Drug: carboplatin; Drug: etoposide; Drug: paclitaxel; Drug: topotecan hydrochloride; Radiation: radiation therapy

INTERVENTIONS:
Biological: filgrastim
Drug: carboplatin
Drug: etoposide
Drug: paclitaxel
Drug: topotecan hydrochloride
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Combining more than one drug and giving them before and with radiation therapy may be an effective treatment for limited-stage small cell lung cancer.

PURPOSE: Phase II trial to study the effectiveness of chemotherapy plus radiation therapy in treating patients who have limited-stage small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the complete response rate to 2 courses of paclitaxel and topotecan followed by consolidation chemoradiotherapy in patients with limited stage small cell lung cancer. II. Determine the toxic effects of this regimen in this patient population. III. Describe the pattern of relapse, documenting carefully the location of relapse with respect to the original disease volume and the radiation treatment field in these patients. IV. Determine the overall and failure free survival of these patients.

OUTLINE: Patients receive topotecan IV on days 1-5 and paclitaxel IV over 3 hours on day 1. Filgrastim (G-CSF) is administered subcutaneously every day starting on day 6 until blood counts recover. The course is repeated once beginning on day 22. After restaging, patients begin thoracic radiotherapy daily, five days per week, for 6-7 weeks. On the same day that radiotherapy begins, patients receive carboplatin IV over 1 hour (day 43) and etoposide IV over 1 hour daily for 3 days (days 43-45). The consolidation chemotherapy is repeated every 21 days for a total of 3 courses. Patients with stable or responding disease undergo prophylactic cranial irradiation. Patients are followed at least every 3 months for 2 years, every 6 months for 3 years, and then at least every year.

PROJECTED ACCRUAL: A total of 70 patients will be accrued for this study within 15-18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically confirmed limited stage small cell lung cancer Includes disease restricted to one hemithorax with regional lymph node metastases, including hilar, ipsilateral and contralateral mediastinal lymph nodes Clinically suspected or confirmed supraclavicular lymph node metastases and pleural effusions that are visible on plain chest radiographs, whether cytologically positive or not, are not eligible Unidimensionally or bidimensionally measurable disease

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Life expectancy: Not specified Hematopoietic: Granulocyte count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin less than 1.5 mg/dL SGOT less than 2 times upper limit of normal (ULN) Renal: Creatinine no greater than ULN Other: Not pregnant or nursing Fertile patients must use effective contraception No concurrent active second malignancy except nonmelanoma skin cancer (i.e., completed therapy and considered to be at less than 30% risk of relapse)

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior chemotherapy for small cell lung cancer No other concurrent chemotherapy Endocrine therapy: No concurrent steroids except for adrenal failure No concurrent hormones except for nondisease related conditions (e.g., insulin for diabetes) No concurrent dexamethasone except for intermittent use as an antiemetic or as an adjunct to prophylactic cranial irradiation Radiotherapy: No prior mediastinal radiotherapy Surgery: Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 1999-03; Primary Completion 2004-06 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
response rate | Up to 5 years
overall survival | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Alan P. Lyss, MD, Study Chair — Missouri Baptist Cancer Center
Locations (48):
- United States (48):
  - Veterans Affairs Medical Center - Birmingham, Birmingham, Alabama
  - University of California San Diego Cancer Center, La Jolla, California
  - UCSF Cancer Center and Cancer Research Institute, San Francisco, California
  - Veterans Affairs Medical Center - San Francisco, San Francisco, California
  - CCOP - Christiana Care Health Services, Wilmington, Delaware
  - Vincent T. Lombardi Cancer Research Center, Georgetown University, Washington D.C., District of Columbia
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - University of Illinois at Chicago Health Sciences Center, Chicago, Illinois
  - Veterans Affairs Medical Center - Chicago (Westside Hospital), Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Veterans Affairs Medical Center - Togus, Togus, Maine
  - Marlene & Stewart Greenebaum Cancer Center, University of Maryland, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - Veterans Affairs Medical Center - Minneapolis, Minneapolis, Minnesota
  - Veterans Affairs Medical Center - Columbia (Truman Memorial), Columbia, Missouri
  - Ellis Fischel Cancer Center - Columbia, Columbia, Missouri
  - Barnes-Jewish Hospital, St Louis, Missouri
  - Missouri Baptist Cancer Center, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Norris Cotton Cancer Center, Lebanon, New Hampshire
  - Veterans Affairs Medical Center - Buffalo, Buffalo, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - CCOP - North Shore University Hospital, Manhasset, New York
  - North Shore University Hospital, Manhasset, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - New York Presbyterian Hospital - Cornell Campus, New York, New York
  - Mount Sinai Medical Center, NY, New York, New York
  - CCOP - Syracuse Hematology-Oncology Associates of Central New York, P.C., Syracuse, New York
  - State University of New York - Upstate Medical University, Syracuse, New York
  - Veterans Affairs Medical Center - Syracuse, Syracuse, New York
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - Veterans Affairs Medical Center - Durham, Durham, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - CCOP - Southeast Cancer Control Consortium, Winston-Salem, North Carolina
  - Comprehensive Cancer Center of Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio
  - Rhode Island Hospital, Providence, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - Veterans Affairs Medical Center - Memphis, Memphis, Tennessee
  - University of Tennessee, Memphis Cancer Center, Memphis, Tennessee
  - Vermont Cancer Center, Burlington, Vermont
  - Veterans Affairs Medical Center - White River Junction, White River Junction, Vermont
  - Veterans Affairs Medical Center - Richmond, Richmond, Virginia
  - MBCCOP - Massey Cancer Center, Richmond, Virginia

REFERENCES:
- [Result] Bogart JA, Herndon JE 2nd, Lyss AP, Watson D, Miller AA, Lee ME, Turrisi AT, Green MR; Cancer and Leukemia Group B study 39808. 70 Gy thoracic radiotherapy is feasible concurrent with chemotherapy for limited-stage small-cell lung cancer: analysis of Cancer and Leukemia Group B study 39808. Int J Radiat Oncol Biol Phys. 2004 Jun 1;59(2):460-8. doi: 10.1016/j.ijrobp.2003.10.021. PMID 15145163
- [Result] Cicchetti MG, Bogart J, Lyss A, et al.: Spinal cord dose in limited stage small cell lung cancer: a preliminary Quality Assurance Review Committee (QARC) report on CALGB 39808, using target thoracic radiotherapy (TRT) doses of 60 - 70 Gy. [Abstract] Int J Radiat Oncol Biol Phys 51(3 suppl 1): A-656, 356, 2001.
- [Result] Lyss AP, Herndon JE, Bogart JE, et al.: Topotecan (Topo) + paclitaxel (Tax) + G-CSF (G) induction followed by concurrent chemoradiotherapy (CCRT) for patients (pts) with limited stage small cell lung cancer (L-SCLC): preliminary analysis of CALGB 39808. [Abstract] Proceedings of the American Society of Clinical Oncology 20: A-1270, 2001.